CLINICAL TRIAL: NCT02932449
Title: A 5-year Longitudinal Observational Study of Patients With Primary Biliary Cholangitis
Status: Completed | Type: Observational
Sponsor: Target PharmaSolutions, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TARGET-PBC
Record Dates: First submitted 2016-09-07; First posted 2016-10-13 (Estimated); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Biliary Cirrhosis, Primary
MeSH Terms: conditions — Liver Cirrhosis, Biliary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Participants enrolled in TARGET-PBC will be invited to participate in the optional Biorepository Specimen Bank (BSB). Blood samples for biomarker and DNA/RNA assays will be collected on a voluntary basis and participation in this project will not affect participation in the main study.
  Blood samples for exploratory genetic and biomarker studies can be used for research purposes to identify potential biomarkers predictive of PBC diagnosis, assess correlates of response to PBC treatment (in terms of mode of action, efficacy, dose, safety and tolerability), understand factors influencing disease progression, determine how best to monitor and treat PBC, aid in the development of a new medical products, or explore complications of PBC and treatment.
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a 5-year, longitudinal, observational study of patients with PBC designed to specifically address important clinical questions that remain incompletely answered from registration trials. In addition to the study database, a bio specimen repository will also be included so that translational studies of genomics and biomarkers of response may be performed.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age 18 or older) being treated or managed for PBC

Exclusion Criteria:

* Inability to provide written informed consent
* Simultaneous enrollment in another prospective registry or clinical trial or study where PBC treatment outcomes are reported, except where approved or conducted as an adjunct project of TARGET-PBC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults with PBC who are being seen specifically to address this disease process
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2016-10; Primary Completion 2025-01-23 (Actual); Study Completion 2025-01-23 (Actual)

PRIMARY OUTCOMES:
Evaluate PBC treatment regimens being used in clinical practice | up to 5 years
Examine populations underrepresented in phase III clinical trials | up to 5 years
Examine biochemical response and its association with long term outcomes | up to 5 years
Estimate adverse event frequency and severity and describe management practices | up to 5 years

CONTACTS AND LOCATIONS:
Locations (39):
- United States (39):
  - Institute for Liver Health, Chandler, Arizona
  - Banner University Medical Center, Phoenix, Arizona
  - Mayo Clinic, Phoenix, Arizona
  - University of Arkansas, Little Rock, Arkansas
  - Stanford University Medical Center, Palo Alto, California
  - California Liver Research Institute, Pasadena, California
  - University of California Davis, Sacramento, California
  - University of Colorado- Anschutz Medical Campus, Aurora, Colorado
  - Yale Internal Medicine, Digestive Diseases, New Haven, Connecticut
  - Gastro Florida, Clearwater, Florida
  - University of Florida Hepatology Research, Gainesville, Florida
  - SCFLD/University of Miami, Miami, Florida
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - Illinois Gastroenterology Group, Arlington Heights, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Mercy Medical Center, GI Research, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Southern Therapy and Advanced Research LLC (STAR), Jackson, Mississippi
  - Saint Louis University, St Louis, Missouri
  - University of Nebraska, Omaha, Nebraska
  - Sandra Atlas Bass Center for Liver Diseases, Manhasset, New York
  - NYU Langone Health, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Center for Liver Disease and Transplant at CMC, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - Baylor,Scott and White All Saints, Fort Worth, Texas
  - Liver Associates of Texas, P.A., Houston, Texas
  - Pinnacle Clinical Research, Live Oak, Texas
  - Bon Secours Liver Institute of Virginia, Richmond, Virginia
  - Virginia Commonwealth University (VCU), Richmond, Virginia
  - University of Washington, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided